CLINICAL TRIAL: NCT01408147
Title: Prevention of Postpartum Weight Retention in Low Income WIC Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Professor-Principal Investigator, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DK087889-01A1 (NIH)
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: Postpartum weight retention; Low income women; WIC; Online
MeSH Terms: conditions — Obesity; Gestational Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): This group will be allowed access to an online weight loss program. The program is designed to help low income women lose weight through lifestyle intervention.
  Interventions: Behavioral: Online postpartum weight control
- Standard WIC care (No Intervention): The control group will received Standard Care as provided through WIC.

INTERVENTIONS:
Behavioral: Online postpartum weight control — The intervention group will be given access to an online weight loss program supplemented by monthly group meetings.
  Other Names: Internet-based treatment for weight loss
  Arms: Treatment Group

SUMMARY:
This study will examine the effects of an online behavioral intervention to promote weight loss in low income postpartum women in the WIC program.

DETAILED DESCRIPTION:
This program is designed to reduce postpartum weight retention in low income women in the WIC program. The weight loss program will be delivered over the internet and will use behavioral weight loss techniques.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-40 years.
* Delivery within 6-52 weeks
* Exceed pre-pregnancy weight by at least 4.5 kg (10 pounds) or current body mass index (BMI) >/= 25
* Current BMI > 22
* English or Spanish speaking
* Has internet access at home or a landline
* Literacy of at least 5th grade reading level
* Has a cell phone

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Relocating in the next year
* Serious psychological problems (untreated depression, schizophrenia, bipolar disorder) or medical problem (i.e. heart disease, cancer, renal disease and diabetes), for which physician supervision of diet and exercise prescription is needed.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 371 (Actual)
Dates: Start 2011-07; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD., Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (2):
- United States (2):
  - California Polytechnic State University, San Luis Obispo, California
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Background] Phelan S, Hagobian T, Brannen A, Hatley KE, Schaffner A, Munoz-Christian K, Tate DF. Effect of an Internet-Based Program on Weight Loss for Low-Income Postpartum Women: A Randomized Clinical Trial. JAMA. 2017 Jun 20;317(23):2381-2391. doi: 10.1001/jama.2017.7119. PMID 28632867
- [Background] Martin CL, Tate DF, Schaffner A, Brannen A, Hatley KE, Diamond M, Munoz-Christian K, Pomeroy J, Sanchez T, Mercado A, Hagobian T, Phelan S. Acculturation Influences Postpartum Eating, Activity, and Weight Retention in Low-Income Hispanic Women. J Womens Health (Larchmt). 2017 Dec;26(12):1333-1339. doi: 10.1089/jwh.2016.6154. Epub 2017 Aug 17. PMID 28816589
- [Result] Phelan S, Brannen A, Erickson K, Diamond M, Schaffner A, Munoz-Christian K, Stewart A, Sanchez T, Rodriguez VC, Ramos DI, McClure L, Stinson C, Tate DF. 'Fit Moms/Mamas Activas' internet-based weight control program with group support to reduce postpartum weight retention in low-income women: study protocol for a randomized controlled trial. Trials. 2015 Feb 25;16:59. doi: 10.1186/s13063-015-0573-9. PMID 25887964
- [Derived] Bennion KA, Tate D, Munoz-Christian K, Phelan S. Impact of an Internet-Based Lifestyle Intervention on Behavioral and Psychosocial Factors During Postpartum Weight Loss. Obesity (Silver Spring). 2020 Oct;28(10):1860-1867. doi: 10.1002/oby.22921. Epub 2020 Sep 4. PMID 32888250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 WIC Clinics Recruited; 371 participants total across all clinics
Units Other Than Participants: 12
Period: Overall Study
Arm/Group | Treatment Group | Standard WIC Care
Started | 174; 5 12 (174 participants) | 197; 6 12 (197 participants)
Completed | 174; 5 12 (1 clinic withdrew due to low census) | 196; 6 12
Not Completed | 0; 0 12 | 1; 0 12
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Across the 11 clinics, 371 participants were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Standard WIC Care | Total
Number analyzed (Participants) | 174 | 197 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (5.2) | 28.6 (5.5) | 28.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 197 | 371
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 146 | 157 | 303
  Not Hispanic or Latino | 28 | 40 | 68
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 174 | 196 | 370

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Women randomized to the weight loss group will be assessed over time at study entry, 6 months, and 12 months.
  The primary outcome is change from entry to the endpoint at 12 months.
Time Frame: 12 months
Population: This cluster randomized trial included 11 clinics. Participant numbers reflect number of people randomized within the clinics.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Treatment Group | Standard WIC Care
Number analyzed (Participants) | 174 | 196
kg | -3.2 [-4.1 to -2.4] | -0.9 [-1.7 to -0.1]
Statistical Analysis 1: Comparison: Treatment Group vs Standard WIC Care; To test the primary hypothesis, a generalized linear mixed effect model was used (intervention group as a fixed effect and clinic and subject as random effects). A group x time interaction term (fixed effect) tested if the change in weight over time differed significantly. The model included participant-level covariates (i.e., ethnicity, weeks postpartum at study entry, lactation, and age); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.3

2. Secondary Outcome: Calorie Intake
Description: Calorie intake was measured over time at study entry, 6 and 12 months. The primary outcome is change from entry to 12 months.
Time Frame: 12 months
Population: 12 clusters were randomized. Sample size above reflect total number of participants in each group.
Measure: Least Squares Mean (95% Confidence Interval); unit: kcal/day
Arm/Group | Treatment Group | Standard WIC Care
Number analyzed (Participants) | 170 | 191
kcal/day | -298 [-423 to -174] | -144 [-257 to -32]

ADVERSE EVENTS:
Arm/Group | Treatment Group | Standard WIC Care
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/196
Other Adverse Events (participants affected / at risk) | 16/174 | 15/196
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=174) | Standard WIC Care (N=196)
Self-reported injury from physical activity (Injury, poisoning and procedural complications) | 16 (16) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No